CLINICAL TRIAL: NCT02089568
Title: Are Prophylactic Antibiotics Necessary Before Laparoscopic Living Kidney Donation? A Double Blind, Randomised, Controlled Trial.
Brief Title: Prophylaxis Of Wound Infections- Antibiotics in Renal Donation
Acronym: POWAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nizam Mamode, Consultant Transplant Surgeon, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POWAR; 2012-000942-36 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Infection
Keywords: Living donation; Antibiotics; Laparoscopic surgery
MeSH Terms: conditions — Infections | interventions — Amoxicillin-Potassium Clavulanate Combination; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: co-amoxiclav (Experimental): experimental
  Interventions: Drug: Co-Amoxiclav
- Control (Placebo Comparator): comparator
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Co-Amoxiclav — Will receive 1.2g co-amoxiclav at induction
  Other Names: Augmentin
  Arms: Drug: co-amoxiclav
Drug: Normal Saline — Placebo - 0.9% saline
  Arms: Control

SUMMARY:
The aim of this study is to see whether antibiotics given at the start of laparoscopic kidney donation surgery prevent infection.

DETAILED DESCRIPTION:
Subjects undergoing laparoscopic donor nephrectomy will be randomised to either a single dose of intravenous co-amoxiclav or placebo prior to surgery. Outcome measures include any infections, length of stay and costs

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (over 18 years) undergoing hand-assisted laparoscopic donor nephrectomy, who have given written informed consent, will be included.
* Patients whose first language is not English will be included; they comprise a significant part of our patient population and we will use translation services as is our normal practice.
* Women of child-bearing age taking adequate contraception will be included.

Exclusion Criteria:

* Patients with a known allergy to penicillin or other antibiotics.
* Patients with MRSA colonisation.
* Participation in another investigational study within the previous 90 days.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rate of infection after surgery | 24 months

SECONDARY OUTCOMES:
Ultrasonic evidence of wound healing | 24 months
  Wounds will be assessed using high resolution ultrasound to assess dermal and epidermal healing.
Length of hospital stay | 24 months
Readmission rates | 24 months
Antibiotic associated side effects | 24 months
  Including diarrhoea and allergic reactions
Return to work and normal activities | 24 months
Quality of life | 24 months
Relative costs | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nizam Mamode, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom